CLINICAL TRIAL: NCT04520152
Title: Evaluation of the Free Flow Medical Lung Tensioning Device System for the Treatment of Severe Emphysema - EFFORT
Brief Title: Evaluation of the Free Flow Medical Lung Tensioning Device System for the Treatment of Severe Emphysema
Acronym: EFFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, Prof. dr. D.J. Slebos MD, PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFFORT
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Emphysema or COPD
Keywords: lung volume reduction; nitinol; device
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Bronchoscopic LTD placement
  Interventions: Device: FreeFlowMedical Lung Tensioning Device

INTERVENTIONS:
Device: FreeFlowMedical Lung Tensioning Device — Bronchoscopic lung tensioning device implantation

SUMMARY:
Patients with severe emphysema have limited options for treatment. Current treatments include lung transplant, lung volume reduction surgery or endobronchial lung volume reduction using valves or coils. These options are only available for a small and selected group of patients. The Free Flow Medical Lung Tensioning Device System (LTD) is thought to be the next generation endobronchial treatment for patients with severe emphysema designed to address this unmet need. The LTD is designed to compress the areas of lung parenchyma most damaged by emphysema and to tension surrounding tissue to help restore lung elastic recoil in a similar manner to the lung volume reduction coils.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD
2. FEV1/FVC ≤ 70%
3. ≥ 40 years of age
4. Post-bronchodilator FEV1 ≤ 45% of predicted
5. Total Lung Capacity > 100% of predicted
6. Residual Volume (RV) > 175% of predicted
7. RV/TLC > 55%
8. Marked dyspnea defined by a score of ≥ 2 on mMRC dyspnea scale of 0-4
9. Emphysema with ≥ 20% destruction (on -950 Hounsfield units) of two potential treatment lobe(s)
10. Stopped smoking for ≥ 6 months prior to entering the study
11. Completed a pulmonary rehabilitation program prior to entering the study and/or have regular (at least once a week) physiotherapy
12. Ability to read, understand and sign the informed consent form

Exclusion Criteria:

1. History of recurrent clinically significant respiratory infections and/or COPD exacerbations, defined as ≥ 2 hospitalizations for respiratory infections and/or COPD exacerbations during the year prior to enrolment
2. History of recurrent clinically significant respiratory infections and/or COPD exacerbations, defined as ≥ 3 courses of prednisolone and/or antibiotics for respiratory infections and/or COPD exacerbations during the year prior to enrolment
3. Clinically significant bronchiectasis
4. Severe gas exchange abnormalities defined by PaCO2 > 7.0 kPa (52 mmHg) and/or PaO2 < 7.0 kPa (52 mmHg) (measured on room air)
5. ≥ 10 mg prednisone (or equivalent dose of other corticosteroids) daily
6. Inability to walk > 140 meters in 6 minutes
7. Known pulmonary hypertension defined by right ventricular systolic pressure > 45 mmHg and/or evidence of pulmonary hypertension of right ventricular failure on echocardiogram
8. Significant paraseptal emphysema
9. Giant bullae (>1/3 of lung volume)
10. Medical history of asthma
11. Underwent previous LVRS, lobectomy, pneumonectomy or lung transplant
12. Underwent previous treatment with thermal vapor ablation, AeriSeal, Cryospray, endobronchial coils or endobronchial valves (if still implanted)
13. Evidence of other disease(s) that have a predicted survival of less than one year
14. Inability to tolerate bronchoscopy under general anaesthesia
15. Maintenance antiplatelet (except aspirin/Ascal) or anticoagulant therapy (such as warfarin, Coumadin, heparin, LMWH, DOACs, etc) which cannot be permanently stopped prior to entering the study
16. Pregnant, lactating or plans to become pregnant within the study timeframe
17. Known sensitivity to drugs required to perform bronchoscopy under general anaesthesia
18. Any other disease, condition(s) or habit(s) that would interfere with completion of study and follow up assessments, would increase risks of bronchoscopy or assessments or in the judgment of the investigator would potentially interfere
19. Known Nickel, Titanium, or Nitinol allergy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Safety: type and frequency of device-related and procedure-related AE | 3 months
  To evaluate the safety of the LTD in COPD patients with heterogeneous and homogeneous emphysema by evaluating the type and frequency of device-related and procedure-related AE experienced during and following LTD placement through the 3-month visit.
Procedural succes | 3 months
  To evaluate the feasibility of the LTD in COPD patients with heterogeneous and homogeneous emphysema by measuring the frequencies of successful and unsuccessful intended LTD placements.

SECONDARY OUTCOMES:
Performance - Quality of Life: St George's Respiratory Questionnaire | 3 months
  Change in St George's Respiratory Questionnaire total score

CONTACTS AND LOCATIONS:
Locations (2):
- Dept. of Pneumology and Critical Care Medicine, Thoraxklinik, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No